CLINICAL TRIAL: NCT04620590
Title: DAPASALT: An Open Label, Phase IV, Mechanistic, Study to Evaluate the Natriuretic Effect of 2-Week Dapagliflozin Treatment in Type 2 Diabetes Mellitus Patients With Impaired Renal Function
Brief Title: Dapagliflozin Treatment in Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emerald Clinical Inc. (Industry)
Collaborators: University Medical Center Groningen (Other); Ground Zero Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCG 20-001; 2020-001247-12 (EudraCT Number); HC6-24-c243179 (Other: Health Canada)
Record Dates: First submitted 2020-11-03; First posted 2020-11-09 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2023-04

CONDITIONS: Diabetes Mellitus, Type 2; Impaired Renal Function
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Renal Insufficiency | interventions — dapagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Arm (Experimental): Patients will receive dapagliflozin 10 mg tablets once daily for 14±1 days.
  Interventions: Drug: Dapagliflozin 10 MG [Farxiga]

INTERVENTIONS:
Drug: Dapagliflozin 10 MG [Farxiga] — Dapagliflozin is a stable, reversible, highly selective, and orally active inhibitor of human renal sodium glucose co-transporter 2 (SGLT2), the major transporter responsible for glucose reabsorption in the kidney. Patients will receive one tablet dapagliflozin 10 mg per day for a total period of 14±1 days. This dose is the recommended dose for monotherapy and for add-on combination therapy with other glucose-lowering medicinal products including insulin to improve glycaemic control in T2DM.

SUMMARY:
Open label, mechanistic, single-arm study to evaluate the natriuretic effect of 2 weeks dapagliflozin treatment in T2DM patients with impaired renal function. It will measure the average change in 24-hr sodium excretion from average Baseline to average values at Day 2 to 4 within the study group. The study will allow for an up to 6-week Screening and Run-in Period, a 2-week Treatment Period and a 5-day Follow-up Period. Patients will consume food from standardized food boxes starting on Day -6 (patients not on insulin) or Day -20 at the earliest (patients on insulin) of the study until Day 18 (inclusive). Eligible patients will receive dapagliflozin 10 mg tablets once daily for 14±1 days starting on Day 1. This will be followed by a Follow-up Period of 5 days.

DETAILED DESCRIPTION:
This is an open label, mechanistic, single-arm study to evaluate the natriuretic effect of 2 weeks dapagliflozin treatment in T2DM patients with impaired renal function. The study population is as described below. The maximum duration of the study will be 62 days including the allowed window periods for the study (±1 day for Visit 7 at Day 13). The study will allow for an up to 6-week Screening and Run-in Period. The Run-in Period should always last 6 days for patients not on insulin but may be up to 20 days (day -20 to day -1) for patients on insulin. Patients on insulin may require a longer Run-in Period in order to be able to adjust their insulin requirements according to the caloric content of the food boxes, if needed. It is recommended to keep the insulin dose stable during the trial, but investigators can change the dose if medically required. However, it is not mandatory for the patient on insulin to use the entire extended Run-in Period. Based on the Investigator's judgement, the Run-in Period may be shortened once each patient (on insulin) has had sufficient time to adapt to the food boxes, and it is determined that the patient's insulin requirement has stabilised sufficiently to continue in the study. The study will then include a 2-week Treatment Period (Day 1 to Day 14) and a 5-day Follow-up Period: Day 15 to Day 19. Patients will consume food from standardised food boxes (with sodium content 150 mmol) starting on Day -6 (patients not on insulin) or Day -20 at the earliest (patients on insulin) of the study until Day 18 (inclusive). Eligible patients will receive dapagliflozin 10 mg tablets once daily for 14±1 days starting on Day 1. This will be followed by a Follow-up Period of 5 days.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study-specific procedures.
* Female and/or male aged between 18 years and less than or equal to 80 years.
* A diagnosis of T2DM with HbA1c ≥6.5% (≥48 mmol/mol) and =11% (<97 mmol/mol); and eGFR (CKD-EPI) between ≥25 and ≤50 mL/min/1.73m2.
* Patient specific optimal antihypertensive dose of an ACEi or ARB (as per Investigator's judgement) for at least 6 weeks prior to Visit 4 (Day 1).
* A stable insulin dosing (intermediate, long-acting, premixed insulin, basal bolus insulin) for the last 12 weeks prior to Visit 4 (Day 1) as judged by the Investigator. Metformin, sulphonylurea, DPP4 inhibitors or any combinations of these agents with or without insulin would be accepted but is not mandatory. If used, stable dose of metformin, sulphonylurea, or DPP4 inhibitors or their combination as anti-diabetic therapy for the last 12 weeks prior to start of treatment with dapagliflozin is required.
* Suitable veins for cannulation or repeated venipuncture.
* Female patients must be 1 year post-menopausal, surgically sterile, or using an acceptable method of contraception (an acceptable method of contraception is defined as a barrier method in conjunction with a spermicide) for the duration of the study (from the time they sign consent) and for 3 months after the last dose of study drug to prevent pregnancy. In addition, oral contraceptives, approved contraceptive implant, long-term injectable contraception, intrauterine device, or tubal ligation are allowed. Oral contraception alone is not acceptable; additional barrier methods in conjunction with spermicide must be used.
* Patient specific optimal antihypertensive dose of an ACEi or ARB (as per Investigator's judgement) for at least 6 weeks prior to Visit 4 (Day 1).
* A stable insulin dosing (intermediate, long-acting, premixed insulin, basal bolus insulin) for the last 12 weeks prior to Visit 4 (Day 1) as judged by the Investigator. Metformin, sulphonylurea, DPP4 inhibitors or any combination of these agents with or without insulin would be accepted but is not mandatory. If used, stable dose of metformin, sulphonylurea, or DPP4 inhibitors or their combination as anti-diabetic therapy for the last 12 weeks prior to start of treatment with dapagliflozin is required.

Exclusion Criteria:

* Previous enrolment in the present study or participation in another clinical study with an investigational product during the last 6 months prior to Screening Visit (Visit 1).
* Involvement in the planning and conduct of the study (applies to both UMCG staff and staff at third party vendor or at investigational sites).
* Hypersensitivity to dapaglifozin, indocyanine green, sodium iodide, or iodine, or patients who have poorly tolerated indocyanine green in the past.
* Pacemaker or other implanted electronic devices.
* Pregnancy.
* Breastfeeding.
* Known clinically significant disease or disorder; or clinically relevant abnormal findings in physical examination, clinical chemistry, haematology and urinalysis; or unstable or rapidly progressing renal disease; other dietary restrictions that would make it difficult for the subject to follow the protocol required diet plan or any other condition or minor medical complaint, which, in the opinion of the investigator, may either put the patient atrisk because of participation in the study, or influence the results, or the patient's ability to participate in the study and comply with study procedures, restrictions and requirements.
* Diagnosis of T1DM.
* Hyperthyroidism or autonomic thyroid adenomas.
* Abnormal vital signs, after 10 minutes supine rest, defined as any opf the following (Visit 1); Systolic blood pressure above 180mmHg; Diastolic blood pressure above 110 mmHg; Pulse less than 50 bpm or greater than 100 bpm.
* Any of the following cardiovascular/vascular within 3 months prior to signing the consent at Visit 1, as assessed by the Investigator: myocardial infarction, cardiac surgery or revascularization (coronary artery bypass graft [CABG]/ percutaneous transluminal coronary angioplasty [PTCA], unstable angina, unstable heart failure, heart failure New York Association Class IV, transient ischemic attack or significant cerebrovascular disease, unstable or previously undiagnosed arrhythmia.
* Patients with severe hepatic impairment (Child-Pugh C).
* Ongoing weight-loss diet (hypocaloric diet) or use of weight-loss agents, unless the diet or treatment has been stopped at least 3 months before Screening Visit, ensuring patients having a stable body weight with no verified body weight variability of greater then 3 kg during the 3 months before Screening Visit.
* Symptoms/complaints suggestive of established neurogenic bladder and/or incomplete bladder emptying.
* History of bladder cancer.
* Non-diabetic kidney disease.
* UACR greater than 1000 mg/g per day at the Screening Visit based on spot urine sample (quantitative assessment).
* Current chronic use of the following medication: glucagon-like peptide receptor agonists or thiazolidinediones, oral glucocorticoids, non-steroidal anti-inflammatory drugs (NSAIDs), immune suppressants, chemotherapeutics, antipsychotics, tricyclic antidepressants (TCAs) and monoamine oxidase inhibitors.
* Receiving immunosuppressive or other immunotherapy for primary or secondary renal disease within 6 months prior to Screening Visit (Visit 1).
* Current treatment or treatment within the last 2 weeks prior to Screening Visit (Visit 1) with mineralocorticoid antagonists (loop or thiazide diuretics are allowed as long as they are used in stable dose for at least 4 weeks prior to screening).
* A metformin dose which is outside the specified dose range for renal impairment according to local guidelines and/or Investigator's judgement.
* Medicinal products and substances that can reduce or increase absorption of indocyanine green; anticonvulsants, bisulphite compounds, haloperidol, heroin, meperidine, metamizol, methadone, morphium, nitrofurantoin, opium alkaloids, phenobarbital, phenylbutazone (reduced absorption), and cyclopropane, probenecid, rifamycin (increased absorption).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2021-04-20 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Change in 24-hr sodium excretion | 24 hours
  To investigate change in 24-hr sodium excretion during dapagliflozin treatment between Baseline (average of Days -3 to -1) and average of Days 2 to 4 within each study group in patients with type 2 diabetes mellitus (T2DM) with impaired renal function.

CONTACTS AND LOCATIONS:
Overall Officials: Hiddo JL Heerspink, Principal Investigator — Investigator
Locations (2):
- CU Anschutz Medical Campus - Clinical Translational Research Center (CTRC), Aurora, Colorado, United States
- David Cherney, CM, PhD, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No